CLINICAL TRIAL: NCT01741688
Title: A Multi-National, Multi-Center Non-Interventional Study in Rheumatoid Arthritis (RA) Patients Treated With Tocilizumab
Brief Title: An Observational Study of Tocilizumab (Actemra) in Participants With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28206
Record Dates: First submitted 2012-11-30; First posted 2012-12-05 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tocilizumab: Participants with moderate to severe rheumatoid arthritis (RA), according to the American College of Rheumatology (ACR) criteria and the Disease Activity Score Based on 28 Joints (DAS28), in whom the attending physician has decided to start treatment with tocilizumab (according to the local label).
  Interventions: Biological: Tocilizumab

INTERVENTIONS:
Biological: Tocilizumab — Tocilizumab was administered according to the local label.
  Other Names: Actemra

SUMMARY:
This observational study evaluates the use and efficacy of intravenous (IV) tocilizumab in routine clinical practice in participants with moderate to severe rheumatoid arthritis. Eligible participants initiated on tocilizumab treatment in accordance with the local label were followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults, >/= 18 years of age
* Moderate to severe rheumatoid arthritis according to the revised (1987) American College of Rheumatology (ACR) criteria
* Participants in whom the treating physician has made the decision to commence tocilizumab treatment (in accordance with the local label); this can include participants who have received tocilizumab treatment within 8 weeks prior to the enrollment visit

Exclusion Criteria:

* Participants who have received tocilizumab more than 8 weeks prior to the enrollment visit
* Participants who have received treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational agent, whichever is longer) before starting treatment with tocilizumab
* History of autoimmune disease or any joint inflammatory disease other than rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with rheumatoid arthritis (RA) initiated on treatment with tocilizumab
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-10-26 (Actual); Primary Completion 2014-03-06 (Actual); Study Completion 2014-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Peru (4):
  - ABK Reuma SRL- Medicentro BioCiencias, Lima
  - Hospital de la Mujer, Lima
  - Clinica San Borja; Servicio De Reumatologia, Lima
  - Clinica El Golf, San Isidro

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab
Started | 16
Completed | 13
Not Completed | 3
Not completed — Lack of insurance coverage | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 55 [33.4 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 2
Region of Enrollment [Number; unit: participants]
  Peru | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants on Tocilizumab at 6 Months After Treatment Initiation
Time Frame: At 6 months
Measure: Number; unit: participants
Groups:
- Cohort: Participants with moderate to severe rheumatoid arthritis (RA), according to the American College of Rheumatology (ACR) criteria and the Disease Activity Score Based on 28 Joints (DAS28), in whom the attending physician has decided to start treatment with tocilizumab (according to the local label).
  Tocilizumab: Tocilizumab was administered according to the local label.
Arm/Group | Cohort
Number analyzed (Participants) | 16
participants | 14

2. Secondary Outcome: Percentage of Participants With Systemic Manifestations of Rheumatoid Arthritis
Description: Systemic manifestation measured by C-reactive protein levels > 3
Time Frame: At baseline
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
percentage of participants | 93.8

3. Secondary Outcome: Percentage of Participants Starting Tocilizumab After Prior and Baseline Disease-Modifying Anti-rheumatic Drugs (DMARDs) Exposure
Description: DMARDs exposure was evaluated for all participants. "Prior DMARDs treatment" includes participants, who were treated with DMARDs 6 months before being included in the study. "DMARDs treatment at baseline" includes participants, who were receiving DMARDs when they were included in the study and continued with this concomitant medication to tocilizumab.
Time Frame: At baseline
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
percentage of participants
  Prior DMARDs treatment | 18.8
  DMARDs treatment at baseline | 62.5

4. Secondary Outcome: Number of Participants Starting Tocilizumab After Failing Other Biologic Agents
Description: Other biologic agents include anti-Tumor Necrosis Factor (TNF) antibody.
Time Frame: At baseline
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
participants | 1

5. Secondary Outcome: Median Dose at 6 Months
Time Frame: At 6 months
Population: Number of participants remaining in the study at 6 months
Measure: Median (Full Range); unit: mg/kg of body weight
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
mg/kg of body weight | 8 [6.3 to 9.2]

6. Secondary Outcome: Number of Participants With Dose Modifications at 6 Months
Time Frame: At 6 months
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 14
participants | 4

7. Secondary Outcome: Median Duration of Treatment
Time Frame: Approximately 16 months
Measure: Median (Full Range); unit: months
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
months | 6 [3.4 to 6.8]

8. Secondary Outcome: Percentage of Participants Discontinued From Tocilizumab for Safety
Description: Safety variable measuring number of patients that discontinued tocilizumab due to adverse reactions to tocilizumab.
Time Frame: Approximately 16 months
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
percentage of participants | 0

9. Secondary Outcome: Percentage of Participants Discontinued From Tocilizumab for Lack of Efficacy
Description: Efficacy variable that measures the rate of participants discontinued from tocilizumab due to lack of efficacy according to criteria of treating physician.
Time Frame: Approximately 16 months
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
percentage of participants | 0

10. Secondary Outcome: Number of Participants Discontinued From Tocilizumab for Other Reasons
Description: This variable measures the number of events not related to safety or efficacy leading to discontinuation of tocilizumab treatment.
Time Frame: Approximately 16 months
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
participants | 3

11. Secondary Outcome: Time to Restoration of Initial Dosing Regimen
Time Frame: Approximately 16 months
Reporting Status: Not Posted

12. Secondary Outcome: Non-adherence Rate of Physician to the Recommended Dosing Regimen
Time Frame: Approximately 16 months
Reporting Status: Not Posted

13. Secondary Outcome: Percentage of Participants on Tocilizumab Monotherapy at Study Entry
Time Frame: At baseline
Measure: Number; unit: percentage of participants
Arm/Group | Cohort
Number analyzed (Participants) | 16
percentage of participants | 12.5

14. Secondary Outcome: Total Tender Joint Count (TJC)
Time Frame: At Visit 1 (Baseline), Observation 1: up to 4 weeks, Observation 2: up to 8 weeks; Observation 3: up to 12 weeks; Observation 4: up to 16 weeks and Observation 5: up to 20 weeks
Measure: Median (Full Range); unit: Number of tender joints/participant
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
Number of tender joints/participant
  Visit 1 | 18 [12 to 22]
  Observation 1 | 0 [0 to 5]
  Observation 2 | 0 [0 to 6]
  Observation 3 | 0 [0 to 0]
  Observation 4 | 0 [0 to 0]
  Observation 5 | 0 [0 to 0]

15. Secondary Outcome: Total Swollen Joint Count (SJC)
Time Frame: as for outcome 14
Measure: Median (Full Range); unit: Number of swollen joints/participant
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
Number of swollen joints/participant
  Visit 1 | 18 [5 to 18]
  Observation 1 | 0.5 [0 to 8]
  Observation 2 | 0 [0 to 6]
  Observation 3 | 0 [0 to 10]
  Observation 4 | 0 [0 to 0]
  Observation 5 | 0 [0 to 0]

16. Secondary Outcome: Disease Activity Score Based on 28 Joints (DAS28)
Description: The DAS28 is a measure of disease activity in rheumatoid arthritis (RA) and the number 28 refers to the 28 joints that are examined in this assessment. To calculate the DAS28 the following assessments are done: 1) count the number of swollen joints (out of the 28 [sw28]), 2) count the number of tender joints (out of the 28 [t28]), 3) measure Erythrocyte Sedimentation Rate (ESR), and 4) ask the participant to make a 'global assessment of health' (GH) indicated by marking a 10 cm line between very good and very bad.
  The Score is developed under the follow formula:
  DAS28(4) = 0.56*sqrt(t28) + 0.28*sqrt(sw28) + 0.70*Ln(ESR) + 0.014*GH Where, t=tender joints; sw=swollen joints; ESR= Erythrocyte Sedimentation Rate; GH=Global assessment of health score.
  This score may range from 0 to 9.3, where a DAS28 of greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission.
Time Frame: as for outcome 14
Measure: Median (Full Range); unit: DAS28 score
Arm/Group | Tocilizumab
Number analyzed (Participants) | 16
DAS28 score
  Visit 1 | 6.29 [4.82 to 6.72]
  Observation 1 | 2.87 [1.89 to 3.67]
  Observation 2 | 2.23 [2.02 to 3.38]
  Observation 3 | 2.16 [1.82 to 2.80]
  Observation 4 | 2.45 [2.45 to 2.45]
  Observation 5 | 2.41 [2.41 to 2.41]

ADVERSE EVENTS:
Time Frame: From baseline to end of study, approximately 16 months.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=16)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=16)
Keratitis (Eye disorders) | 1 (1)
Corneal ulcer (Eye disorders) | 1 (1)
Flu (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.